CLINICAL TRIAL: NCT04910646
Title: The Evaluation of Orange Peel Fermentation on Body Fat Lowering Efficacy in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201912030RSA
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Fat-lowering

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orange peel fermentation (Experimental)
  Interventions: Drug: orange peel fermentation
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: orange peel fermentation — To evaluate whether the fermented orange peel enzyme has the effect of reducing body fat.
  Arms: orange peel fermentation
Drug: Placebo — Placebo without orange peel fermentation
  Arms: placebo

SUMMARY:
Overweight and obesity can lead to the occurrence of many chronic diseases. In addition to the body mass value (BMI), the excess body fat can also be used as criteria for assessing obesity. Citrus peels are rich in many substances including limonene, Nobiletin, 3-methoxynobiletin, and flavonoids. They could be used for lowering blood pressure and reducing blood pressure, anti-anxiety and sleep aid and etc. Fermentation technology is used to ferment the peel to increase the content of neutral components in citrus peel. Therefore, I want to evaluate whether the fermented orange peel enzyme has the effect of reducing fat.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 20 and 65 who are willing to sign the consent form of the subject.
2. For those with BMI ≥ 24 or fatty liver, men's body fat ≥ 25%, women's body fat ≥ 30%
3. Those who are not pregnant and are willing to cooperate with contraception during the trial period.
4. Those who have no history of cardiovascular disease, organ transplantation, epilepsy or convulsions, liver and kidney disease, malignant tumors, endocrine disease, mental disease, alcohol or drug abuse, and other major organic diseases (according to medical history).

Exclusion Criteria:

1. Pregnant women, people with a history of cardiovascular disease, organ transplantation, epilepsy or convulsions, liver and kidney disease, malignant tumors, endocrine diseases, mental illness, alcohol or drug abuse, and other major organic diseases (according to medical history).
2. Those who had undergone major surgery or bariatric surgery (according to medical history).
3. Currently or within 3 months before participating in the screening, those subjects used drugs that can affect body fat or increase weight significantly, such as systemic corticosteroids, tricyclic antidepressants, atypical psychiatric drugs, and mood stability Drugs (according to medical history) will be excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2024-06-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether the fermented orange peel enzyme has the effect of reducing fat. | 8 weeks
  Obesity related markers